CLINICAL TRIAL: NCT04190277
Title: Safety Assessment of DBLUS System in Adolescent and Adult Patients With Type 1 Diabetes and Assessment of Its Clinical Efficacy in a Randomized Trial for 3 Months Followed by an Extension Period
Brief Title: Safety Assessment of DBLUS System in Adolescent and Adult Patients With Type 1 Diabetes and Assessment of Its Clinical Efficacy (DIABELOOP SP8)
Acronym: DIABELOOP SP8
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-A01975-52
Record Dates: First submitted 2019-11-19; First posted 2019-12-09 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 1; Closed-Loop
Keywords: Artificial Pancreas; Adolescents; Adults
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 36-week Closed-Loop (Experimental): 2-week baseline period in open-loop condition, then 12-week period in closed-loop condition followed by a 24-week extension period in closed-loop condition
  Interventions: Device: Open-loop condition; Device: Closed-loop condition
- 12-week open-loop and 24-week closed-loop (Active Comparator): 2-week baseline period in open-loop condition, then 12-week period in open-loop condition followed by a 24-week extension period in closed-loop condition
  Interventions: Device: Open-loop condition; Device: Closed-loop condition

INTERVENTIONS:
Device: Open-loop condition — Patient's standard insulin pump setting combined with continuous glucose monitoring sensor
Device: Closed-loop condition — Closed-loop algorithm system paired with continuous glucose monitoring sensor

SUMMARY:
This clinical trial is a randomized trial including a 3-month single-arm part and a 6-month extension phase.

* Following randomization between the 1st group and 2nd group, a 2-week baseline period in open-loop for 148 adults and 30 adolescents will be performed. Patients will receive the standard of care treatment including their usual subcutaneous insulin pump augmented with continuous glucose measurement with Dexcom G6.
* Then, a 3-month study phase will be performed during 12 weeks:

  * 1st group (111 adults randomized from 148 adults and 30 adolescents) will receive the treatment via the Closed-loop System (closed-loop condition).
  * 2nd group (37 adult controls randomized from 148 adults) will receive the standard of care treatment including their usual subcutaneous insulin pump augmented with continuous glucose measurement with Dexcom G6 (open loop condition).
* An extension period of 6 months with the Closed-loop System (closed-loop condition) will be performed at the end of the study phase for all patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* age 14 - 75 years at time of screening
* Type 1 diabetes
* Subject has a clinical diagnosis of type 1 diabetes for at least 2 years as determined via medical records or source documentation by an individual qualiﬁed to make a medical diagnosis.
* An insulin pump user for at least 6 months (with or without CGM experience),
* Living in an area covered by a GSM (Global System for Mobile Communications) network
* Patient not isolated, does not live alone, or has a person living nearby who has a telephone and a key to his or her home
* Patient willing to wear the system continuously throughout the study
* Has TSH in the normal range
* if subject has celiac disease, it has been adequately treated as determined by the investigator
* With history of cardiovascular event 1 year or more from the time of screening must have an EKG within 6 months prior to screening and a stress test within 6 months prior to screening or during screening. If subject has an abnormal stress test, he will not be allowed to participate in the study, unless there is clearance from a cardiologist. If subject fails stress test, participation is allowed only if there is clearance from a cardiologist
* With 3 or more cardiovascular risk factors listed below must have an EKG within 6 months prior to screening or during screening. If subject has an abnormal EKG, participation is allowed if there is clearance from a cardiologist. Cardiovascular risk factors include:

  * Age >35 years
  * Type 1 diabetes of >15 years' duration
  * Presence of any additional risk factor for coronary artery disease
  * Presence of microvascular disease (proliferative retinopathy or nephropathy, including microalbuminuria)
  * Presence of peripheral vascular disease
  * Presence of autonomic neuropathy
* Must be able to speak and be literate in French
* For adults (18 - 75 years old): having provided written informed consent
* For adolescents (14 - 17 years old): having provided written assent & parents/guardian having provided written informed consent

Exclusion Criteria:

* Patient receiving a total daily dose of insulin lower than 8 U
* Patient with a daily dose of insulin required greater than 90 units
* Patient having severe problems of uncorrected hearing and/or visual acuity
* Patient unable to understand and perform all of the instructions provided by Diabeloop SA
* Subject is unable to tolerate tape adhesive around the sensor or pump placements
* Has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection)
* Has had any of the following cardiovascular events within 1 year of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
* Is being treated for hyperthyroidism at time of screening
* Has diagnosis of adrenal insufficiency
* Has taken any oral, injectable, or intravenous (IV) steroids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV steroids during the study
* Females who are sexually active and able to conceive will be excluded if they are not using an effective method of contraception and do not agree to continue using an effective method of contraception for the duration of the study as determined by investigator.
* Actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks
* Currently abusing illicit drugs
* Currently abusing marijuana
* Currently abusing prescription drugs
* Currently abusing alcohol
* Subject is using pramlintide (Symlin), DDP-4 inhibitor, liraglutide (Victoza or other GLP-1 agonists), metformin, canagliflozin (Invokana or other SGLT2 inhibitors) at time of screening
* Subject has elective surgery planned that requires general anesthesia during the study
* Has a sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening
* Plans to receive red blood cell transfusion or erythropoietin over study participation
* Diagnosed with current eating disorder such as anorexia or bulimia
* Diagnosed with chronic kidney disease that results in chronic anemia
* Hematocrit that is below the normal reference range of lab used
* Patient who has had a pancreatectomy or who has pancreatic malfunctions
* Patient with pancreatic islet transplantation or pancreas transplantation
* Patient on dialysis
* Patient with impaired hepatic functions
* Serum creatinine > 176 µmol/L
* Any other physical or psychological disease, or medication likely to interfere with the conduct of the study and interpretation of the study results as judged by the investigator.
* Pregnancy

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Incidence rate of Serious Adverse Device Effect occuring during the 12-week closed-loop period | 12-weeks closed-loop period
Percentage of time spent in hypoglycemia (glucose level below 70mg/dL (3.9 mmol/L)) between baseline period (2-week period) and in-home study phase in closed-loop (12-week period) for the whole patients of the "single-arm" part | 14-week baseline & closed-loop period
  as recorded by continuous subcutaneous glucose monitoring (CGM)
Difference in percentage of time spent in hypoglycemia (<70mg/dL) during 12 weeks between closed-loop and open-loop | 12-week period
  as recorded by continuous subcutaneous glucose monitoring (CGM)

SECONDARY OUTCOMES:
Percentage of sensor time in glucose level o < 50mg/dL (2.8 mmol/L) o < 60 mg/dL (3.3 mmol/L) o < 70mg/dL (3.9 mmol/L) | during nights, for 24 hours (12:00am-12:00am) and during the following periods: from 12:00am to 6:00am, from 6:00am to 12:00am throughout the 38-week study
  measured by the Dexcom G6 CGM
Number of hypoglycemic episodes with beginning and end of episode o < 70 mg/dL (3.9 mmol/L) o ≤ 54 mg/dL (3 mmol/L) | 36-week period
  as measured by the Dexcom G6 CGM
Incidence of severe hypoglycemia: o Number of severe hypoglycemic episodes needing a third-party intervention o Number of severe hypoglycemic episodes with loss of consciousness o Number of hospitalizations because of a severe hypoglycemia episode | 36-week period
Number of severe hyperglycemia episodes with beginning and end of episode : o > 350 mg/dL (19.4 mmol/L) o > 360 mg/dL (20 mmol/L) or significant ketosis (plasmatic ketones > 3 mmol/L) as defined by the ADA. | 36-week period
  as measured by the Dexcom G6 CGM
Incidence of severe hyperglycemia: o Number of hospitalizations because of ketoacidosis (i.e. incidence of DKA) | 36-week period
Number of technical incidents leading to the interruption of the closed loop | 36-week period
Number of serious adverse events, serious adverse device events, unanticipated adverse device effects | 36-week period
Area under the curve (AUC) from CGM analysis | 36-week period
Risk of hypoglycemia and hyperglycemia (LBGI/HBGI) | 36-week period
  Low Blood Glucose Interstitial & High Blood Glucose Interstitial as measured by the Dexcom G6 CGM
Percentage of time spent in the 70-180 mg/dL target range | during 12 weeks during nights, for 24 hours (12:00am-12:00am) and during the following periods: from 12:00am to 6:00am, from 6:00am to 12:00am throughout the 38-week study
  as recorded by continuous subcutaneous glucose monitoring (CGM)
Percentage of time spent in the 70-180 mg/dL target range | during nights, for 24 hours (12:00am-12:00am) and during the following periods: from 12:00am to 6:00am, from 6:00am to 12:00am throughout the 38-week study
  as recorded by continuous subcutaneous glucose monitoring (CGM)
Percentage of sensor time in glucose level : o < 50 mg/dL (2.8 mmol/L), o < 54 mg/dL (3.0 mmol/L) o < 60 mg/dL (3.3 mmol/L), o < 70 mg/dL (3.9 mmol/L) | during nights, for 24 hours (12:00am-12:00am) and during the following periods: from 12:00am to 6:00am, from 6:00am to 12:00am throughout the 38-week study
  as recorded by continuous subcutaneous glucose monitoring (CGM)
Percentage of sensor time in glucose range 54-70 mg/dL (3.0 - 3.9 mmol/L) | during nights, for 24 hours (12:00am-12:00am) and during the following periods: from 12:00am to 6:00am, from 6:00am to 12:00am throughout the 38-week study
  as recorded by continuous subcutaneous glucose monitoring (CGM)
Percentage of sensor time in glucose range 70-140 mg/dL (3.9 - 7.8 mmol/L) | during nights, for 24 hours (12:00am-12:00am) and during the following periods: from 12:00am to 6:00am, from 6:00am to 12:00am throughout the 38-week study
  as recorded by continuous subcutaneous glucose monitoring (CGM)
Percentage of sensor time in glucose level o > 180 mg/dL (10.0 mmol/L), o > 250 mg/dL (13.9 mmol/L), o > 300 mg/dL (16.7 mmol/L) o > 350 mg/dL (19.4 mmol/L) | during nights, for 24 hours (12:00am-12:00am) and during the following periods: from 12:00am to 6:00am, from 6:00am to 12:00am throughout the 38-week study
  as recorded by continuous subcutaneous glucose monitoring (CGM)
Evolution of glycosylated hemoglobin between inclusion and end of study | at inclusion, after 12-week period, after 24-week extension period
  calculated from CGM data and measured by blood sampling
Average glycemia level during the entire period | 36-week period
  as measured by the Dexcom G6 CGM
Average fasting glycemia level at 6:00 am | 36-week period
  as measured by the Dexcom G6 CGM
Variability of the glycemia level measured by o the glycemic variation coefficient (CV) intra patient: • CV < 36% • CV ≥ 36% o Standard deviation (SD) | 36-week period
Average dose of insulin used & its daily evolution during the entire study duration | 36-week period
Evolution over time of the DBLUS system's performance on a day-to-day and determination of the optimization delay of glycemic control | 36-week period
Percentage of time spent in closed loop mode (i.e. DBLUS System with loop mode operating) | 36-week period
Percentage of time spent in operating mode for the Dexcom G6 CGM | 36-week period
Scoring of the Diabetes Treatment Satisfaction Questionnaire (DTSQ) to evaluate the acceptance | after baseline period (2-week); after12-week-period; after 24-week extension period
Scoring of the Diabetes Quality of Life (DQOL) questionnaire to evaluate the acceptance | after baseline period (2-week); after12-week-period; after 24-week extension period
Scoring of the Hypoglycemia Fear Survey (HFS) questionnaire to evaluate the acceptance | after baseline period (2-week); after12-week-period; after 24-week extension period
Evolution of the weekly average number of CHO intake (for patient with closed-loop) | 36-week period
Questionnaire of usability (for 50 subjects from Arm 1, including 15 adolescents and 35 adults) | after 4 weeks of closed-loop; after 12 weeks of closed-loop

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia FRANC, Dr, Principal Investigator — Sud Francilien Hospital, Corbeil-Essonnes
Locations (9):
- France (9):
  - Caen University Hospital, Caen
  - Sud Francilien Hospital, Corbeil-Essonnes
  - Grenoble University Hospital, Grenoble
  - Marseille - La Conception University Hospital, Marseille
  - Necker-Enfants Malades University Hospital, Paris
  - Reims University Hospital, Reims
  - Strasbourg University Hospital, Strasbourg
  - Toulouse - Purpan University Hospital, Toulouse
  - Toulouse - Rangueil University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franc S, Reznik Y, Amadou C, Penfornis A, Schaepelynck P, Hanaire H, Delemer B, Le Tallec C, Beltrand J, Jeandidier N, Bensaid S, Orlando L, Hannaert P, Benhamou PY, Charpentier G. Safety and glycemic outcomes of DBLG1 coupled to the DANA-i pump in adults and adolescents with type 1 diabetes mellitus. The SP8 trial. J Endocrinol Invest. 2025 Dec 26. doi: 10.1007/s40618-025-02780-5. Online ahead of print. PMID 41452442